CLINICAL TRIAL: NCT01208337
Title: Pharmacodynamics, Pharmacogenomics, and Preliminary Safety and Efficacy of Alemtuzumab Induction and Tacrolimus in Pediatric Intestinal Transplantation (IND # 100496)
Brief Title: Safety and Efficacy of Alemtuzumab in Pediatric Intestinal Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rakesh Sindhi, Professor of Surgery, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB0701088
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2016-06-20 (Estimated); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Evidence of Liver Transplantation; Rejection; ALEMTUZUMAB
Keywords: Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab induction (Other): Intestine transplant recipients who receive induction with alemtuzumab prior to transplantation.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab is a monoclonal antibody directed against the CD52 antigen. A single dose of 0.3-0.4 mg/kg is given to enrolled subjects at the time of intestine transplantation, 30 minutes after premedication with acetaminophen, diphenhydramine and methylprednisolone
  Other Names: Campath H-1 (Genzyme, Cambridge, MA)

SUMMARY:
This open-label clinical trial will evaluate the safety and efficacy of Alemtuzumab (Campath, Bayer Corp., Pittsburgh) in children (0-17) and adults (18-25) receiving intestinal transplant. Seventy-five subjects receiving primary or repeat intestine transplantation will be enrolled. Primary endpoints include the incidence and severity of biopsy-proven acute cellular rejection, the incidence of freedom from steroids at 5 years, and the incidence of subjects with steroid-free Tacrolimus at whole blood concentrations < 10 ng/ml. Secondary endpoints include a) incidence and severity of opportunistic infections (CMV and EBV), post-transplant lymphoproliferative disorder (PTLD), and chronic rejection b) use of non-immunosuppressive co-medications, c) time to repopulation of all lymphocyte subsets, d) longitudinal characterization of donor-specific alloreactivity in mixed lymphocyte responses (MLR), to identify the time at which it decreases to a level less than third-party-specific alloreactivity e) longitudinal expression (mRNA) of genes, to identify rejection- and non-rejection-specific genes and f) characterization of whole genome mutations, which show differences in parent-to-child transmission between rejectors and non-rejectors. This will identify rejection- and non-rejection-specific genes bearing genetic variants, which might impact on gene function, and complement candidate gene identification efforts based on SNP transmission.

DETAILED DESCRIPTION:
Intraoperatively, it is our impression that Alemtuzumab may predispose to mild coagulopathy. Therefore, we have elected to administer steroids, and withhold Alemtuzumab in the operating room for all small bowel transplant recipients.

1. Premedication with acetaminophen 10 mg/kg orally + diphenhydramine 1 mg/kg intravenously + methylprednisolone 2 mg/kg, intravenously will occur 30 minutes before Alemtuzumab administration.
2. Steroids up to 10 mg/kg as bolus will be administered intravenously in the operating room prior to reperfusion of the allograft followed by decreasing amounts of low-dose steroids post-transplant.

   Day 1 post-transplant: up to 5 mg/kg can be given Day 2 post-transplant: up to 4 mg/kg can be given Day 3 post-transplant: up to 3 mg/kg can be given Day 4 post-transplant: up to 2 mg/kg can be given Day 5 post-transplant: up to 1 mg/kg can be given

   Maintenance steroids are tapered thereafter by switching to equivalent amounts of oral prednisone, as soon as ileus results and oral intake intake is possible. By the end of the first month, all patients receive no more than 2.5-5 mg/day of prednisone. This amount is exceeded only if rejection occurs. Long-term prednisone usage may be elected in patients re-transplanted for chronic rejection.
3. A single dose of Alemtuzumab 0.4-0.5 mg/kg will be given intravenously slowly post-operatively. Total dose will not exceed 30 mg.

Procedures:

1. Tacrolimus will be initiated at 0.01 mg per kg body weight orally. If biopsy-proven rejection does not occur, Tacrolimus will be titrated to whole blood concentrations:

   Month 1: 15-20 ng/ml Months 2-3: 10-15 ng/ml Month 4-6: 8-10 ng/ml Months 6-12: 5-10 ng/ml
2. This minimization protocol will be delayed by 3 months if biopsy proven acute cellular rejection occurs. At the event of rejection, Tacrolimus minimization and steroids sparing will be discontinued and standard immunosuppression will be instituted. For example, if rejection occurs, Tacrolimus is increased to month 1 levels of 15-20 ng/ml, and steroids added to the regimen. Steroids will be reduced or eliminated within 3 months of rejection, and tacrolimus minimization resumed as described above. These levels of Tacrolimus are our standards of care in the event of rejection. Current immunosuppressive protocols at our center include rabbit anti-human thymocyte globulin (rATG) with Tacrolimus monotherapy, or Tacrolimus + steroid without induction.
3. Laboratory tests per clinical protocol. The clinical standard of care will be followed in performing post-Tx monitoring labs consisting of complete blood count with differential count, serum sodium, potassium, chloride, bicarbonate, BUN, creatinine and glucose, and liver function tests consisting of Total bilirubin, aspartate alanine transaminase (ALT), aspartate glutamine transaminase (AST), and glutamyl galactosyl transaminase (GGT), and TAC whole blood concentrations. These laboratory tests are performed at least weekly in the first and second months, twice monthly in month 3, and monthly thereafter to the sixth month. The extra 1 to 11 ml needed for pharmacodynamic and pharmacogenomic studies is discussed further in items 5 and in Table 1.
4. Surveillance intestinal allograft biopsies will be performed per clinical surveillance protocol-twice weekly in the first month, weekly in the second month, two-weekly in the third month, and at least monthly thereafter until the end of the 6th month, and at least annually thereafter. Surveillance biopsies are done because no blood test exists to indicate intestinal allograft dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-25 years
* male and female
* Primary intestine transplantation, repeat intestine transplantation, and intestine transplantation in the setting of a previous or simultaneous liver transplantation

Exclusion Criteria:

* documented non-compliance
* known hypersensitivity to egg protein
* pregnancy
* malignancy
* hepatitis C and B defined as anti-HCV antibody positive, and anti-Hepatitis B surface antigen or Hepatitis B core antibody positive or HBV DNA positive.

Ages: 4 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2007-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sindhi, MD, Principal Investigator — Children's Hospital of Pittsburgh of UPMC/University of Pittsburgh

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alemtuzumab Induction
Started | 23
One-year Follow-up | 23
Five-year Follow-up | 20
Completed | 20
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Alemtuzumab Induction
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 5.7 [0.75 to 20.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Primary Isolated Intestine Transplant [Number; unit: participants] | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post Transplant Lymphoproliferative Disorder (PTLD)
Description: Asses safety of Alemtuzumab in combination with Tacrolimus and steroids in twenty-three pediatric intestine allograft recipients by calculating the rate in which PTLD occurred amongst the study population.
Time Frame: 5 Year
Population: Alemtuzumab induction at the time of transplant may reduce the rate of early acute cellular rejection compared with historical controls, but may increase rate of alternate post-transplant complications, such as Post Transplant Lymphoproliferative Disorder (PTLD).
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Induction
Number analyzed (Participants) | 23
participants | 6

2. Secondary Outcome: Incidence of Biopsy-proven Acute Cellular Rejection
Description: Biopsy-proven incidence of acute cellular rejection
Time Frame: 1 Year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Induction
Number analyzed (Participants) | 23
participants | 12

3. Secondary Outcome: Incidence of Patients in Whom Steroids Are Not Used
Description: As part of analysis for assessing effectiveness and safety of Alemtuzumab Induction at the time of transplant, it is important to assess the incidence in which patients enrolled were able to wean off of steroids post-transplant compared to historical controls.
Time Frame: 1 year
Population: Induction of Alemtuzumab at time of transplant may increase the likelihood of weaning off steroids sooner after transplant than patients who did not receive Alemtuzumab as induction immunosuppression medication.
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Induction
Number analyzed (Participants) | 21
participants | 5

4. Secondary Outcome: Incidence of Patients in Whom Tacrolimus Whole Blood Concentration Less Than 10 ng/ml Are Being Used at 1-year Follow-up.
Description: Tacrolimus whole blood concentrations less than 10 ng/ml
Time Frame: 1 year
Population: It is believed that patients whom received Alemtuzumab at the time of transplant and continue post-transplant with functioning grafts will have Tacrolimus whole blood concentrations less than 10ng/ml.
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Induction
Number analyzed (Participants) | 21
participants | 16

5. Secondary Outcome: Incidence of Patients in Whom Steroids Are Not Used
Description: as for outcome 3
Time Frame: 5 year
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Alemtuzumab Induction
Number analyzed (Participants) | 21
participants | 9

ADVERSE EVENTS:
Time Frame: 5 years from time of enrollment
Arm/Group | Alemtuzumab Induction
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alemtuzumab Induction (N=23)
PTLD (Infections and infestations) | 6 (6) — Six of 23 (26%) developed PTLD, including one with Burkitt's lymphoma. These are expected complications of immunosuppression. The incidence was higher than expected from historical incidence of 10-15%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes